CLINICAL TRIAL: NCT01354210
Title: Text Messaging Intervention to Improve ART Adherence Among HIV-positive Youth
Acronym: TXTXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Robert Garofalo, MD, Division Chief - Adolescent Medicine; Director - Center for Gender, Sexuality and HIV Prevention, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: R34DA031053 (NIH); R34DA031053 (NIH)
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Patient Adherence; HIV
Keywords: Patient Adherence; HIV
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care only (No Intervention): The SOC for ART adherence consists of viewing a 20-minute animated tutorial which explains the importance of adherence to antiretroviral medication. It is specifically designed for viewers who have no science background and is appropriate for adolescents and young adults.
- Intervention (Experimental): This study will test a tailored, personalized SMS Text Message Reminder intervention to improve adherence to ART among non-adherent YLH. Participants will use their own cell phones for receipt of the intervention. Participants will have the option to choose a tailored personalized message that may be changed as requested throughout the study period (six months). Taking advantage of the Intelecare technology, participants will be asked to send a text message response indicating that that have successfully (or not) taken their meds per schedule. No identifying patient information will be included in the SMS text to protect patient confidentiality.
  Interventions: Behavioral: SMS Text Message Reminder

INTERVENTIONS:
Behavioral: SMS Text Message Reminder — Daily
  Arms: Intervention

SUMMARY:
The purpose of the proposed study is to test SMS (short message service) text messaging technology to improve medication adherence among youth living with HIV (YLH). The proposed study is a randomized controlled trial of the effect of text message reminders on ART (anti-retroviral therapy) adherence among non-adherent YLH. Daily text message reminders will be sent to patients randomized to the intervention group according to their medication schedule, for 6 months. The investigators will enroll non-adherent YLH, ages 16-29. Half of the sample, randomized to the intervention, will receive daily SMS text message medication reminders and half will be randomized to the control condition and receive standard of care (SOC) only. For the controlled trial, adherence levels and viral load will be collected at baseline, 3-month and 6-month follow-up. In addition, at the end of the initial 6-month enrollment period, participants in the control condition will cross-over to the SMS intervention and participants in the intervention condition will cease to receive the SMS intervention. Adherence and viral load data will be collected from each group at 9- and 12-month follow-up points. The investigators hypothesize that youth in the intervention condition will demonstrate a clinically meaningful increase in adherence at 3 and 6 months post-baseline, from approximately 70% to 90% adherence to ART.

DETAILED DESCRIPTION:
The purpose of the proposed study is to test an intervention using SMS text messaging technology to improve medication adherence among YLH. The proposed study is a randomized controlled trial of the effect of text message reminders on ART adherence rates among non-adherent YLH. Daily text message reminders will be sent to all patients randomized to the intervention group according to their medication schedule, for six months. Participants will have the option to choose a tailored personalized message that may be changed as requested throughout the study period. The investigators will enroll YLH, ages 16-29 (i.e., perinatally, transfusion, or behaviorally acquired -- consistent with our feasibility study and the distribution of infection mode in the primary clinic sites) who have demonstrated poor adherence to ART. Half of the sample, randomized to the intervention, will receive daily short message service (SMS; aka "text message") medication reminders and half will be randomized to the control condition and receive standard of care (SOC) only. For the controlled trial, adherence levels and viral load will be collected at baseline, 3-month and 6-month follow-up. In addition, at the end of the initial 6-month enrollment period, participants in the control condition will cross-over to the SMS intervention for 6 months and participants in the intervention condition will cease to receive the SMS intervention. Adherence and viral load data will be collected from each group at the 9-month and 12-month follow-up points. The advantages of these additional features are that they allow the investigators to offer the intervention to all participants, to evaluate the intervention effect in the control group (to confirm the intervention effect) and to assess sustained intervention effects in the intervention group (post-intervention). Specific Aims:

1. To determine the efficacy of an SMS text messaging intervention on our primary outcome: adherence to ART among poorly adherent YLH, ages 16-29 (a group shown to be at high risk for substance use) over a 6-month intervention period, with effects assessed at 3 and 6-months post-baseline.
2. To explore the efficacy of an SMS text messaging intervention on a secondary, exploratory outcome: viral load and cluster of differentiation 4 (CD4) counts, over a 6-month intervention period, with effects assessed at 3 and 6-months post-baseline.
3. To assess the feasibility, acceptability, and satisfaction of this intervention and clinical trial approach by both objective (e.g., automated message delivery and response counts) and subjective measures (e.g., reported satisfaction, acceptability).

Primary Hypotheses:

1. Youth randomized to the SMS text messaging intervention will show greater improvements in levels of adherence to ART and secondary outcomes during the intervention period at 3 and 6 months post-baseline, in comparison to those receiving standard of care only. The investigators hypothesize at least a 10-point difference in adherence level between groups at 3 and 6 months for the intervention to be clinically meaningful.
2. Youth randomized to SMS text messaging intervention will maintain improvements in adherence (i.e., > 90% adherence) at 9-month and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HIV infection (perinatally, transfusion, or behaviorally acquired; documented by medical record review or verification from referring professional)
* Have cell phone access
* Report regular use of text messaging technology
* 16 to 29 years old
* English-speaking
* On an ART regimen for at least one month at the time of enrollment (i.e., not new to ART) with poor adherence to their antiretroviral regimen. For the purposes of this study, poor adherence will be defined at screening by one or more of the following: a) per the AIDS Clinical Trials Group (ACTG) screening questionnaire, participant reports missing at least one dose in the last week or b) reports missing more than 3 medication doses in the last month.

Exclusion Criteria:

* Do not report regular follow-up with their physician (at least every 3 months)
* Pregnant and on ART only due to pregnancy (i.e., will no longer be prescribed ART after delivery)
* Unable to provide assent or consent.

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Adherence to ART via report on visual analogue scale | prior 30 days
  Adherence to ART via report on visual analogue scale

SECONDARY OUTCOMES:
Viral load | 3-month
  The most recent viral load data will be abstracted from medical records at each time point in RNA copies per milliliter of blood plasma. In addition, as a secondary measure of disease status, CD4 count will also be recorded at each time point in CD4 cells per milliliter of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Garofalo, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois, United States

REFERENCES:
- [Result] Garofalo R, Kuhns LM, Hotton A, Johnson A, Muldoon A, Rice D. A Randomized Controlled Trial of Personalized Text Message Reminders to Promote Medication Adherence Among HIV-Positive Adolescents and Young Adults. AIDS Behav. 2016 May;20(5):1049-59. doi: 10.1007/s10461-015-1192-x. PMID 26362167
- See also: Related Info — http://www.luriechildrens.org